CLINICAL TRIAL: NCT03404271
Title: Time-Restricted Feeding Plus Resistance Training in Active Females: Effects on Body Composition, Muscular Performance and Physiological Variables
Brief Title: Time-Restricted Feeding Plus Resistance Training in Active Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: Metabolic Technologies Inc. (Industry); Dymatize Enterprises, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: 2017-912
Record Dates: First submitted 2018-01-04; First posted 2018-01-19 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Healthy Active Females
MeSH Terms: interventions — beta-hydroxyisovaleric acid; Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Investigators and participants will be blinded to dietary supplement (i.e. HMB or placebo). However, neither the investigators nor participants will be blinded to dietary intervention (TRF or ND) due to the nature of these dietary programs. When possible, outcome assessors will be blinded to group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal Diet (Placebo Comparator): Participants in the normal diet (ND) group will follow a traditional dietary pattern, consisting of eating breakfast and continuing to eat throughout the day until the evening. Participants in this group will receive placebo capsules. Participants in all groups will follow an identical resistance training program and be provided with whey protein supplements.
  Interventions: Other: Resistance Training; Dietary Supplement: Protein Supplementation
- Time-Restricted Feeding (Experimental): Participants in the time-restricted feeding (TRF) group will consume all calories within an 8-hour period of time each day. Participants in this group will receive placebo capsules. Participants in all groups will follow an identical resistance training program and be provided with whey protein supplements.
  Interventions: Other: Resistance Training; Dietary Supplement: Protein Supplementation; Behavioral: Time-Restricted Feeding
- Time-Restricted Feeding plus HMB (Experimental): Participants in the time-restricted feeding plus HMB (TRF+HMB) group will consume all calories within an 8-hour period of time each day. Participants in this group will receive HMB capsules. Participants in all groups will follow an identical resistance training program and be provided with whey protein supplements.
  Interventions: Dietary Supplement: Beta-hydroxy beta-methylbutyrate; Other: Resistance Training; Dietary Supplement: Protein Supplementation; Behavioral: Time-Restricted Feeding

INTERVENTIONS:
Dietary Supplement: Beta-hydroxy beta-methylbutyrate — 3 grams per day of the calcium salt form of beta-hydroxy beta-methylbutyrate (HMB).
  Other Names: HMB
  Arms: Time-Restricted Feeding plus HMB
Other: Resistance Training — Performing supervised resistance training three times per week.
Dietary Supplement: Protein Supplementation — Consuming a protein supplement daily.
Behavioral: Time-Restricted Feeding — Consuming all calories within a specified 8-hour period of time each day.
  Other Names: Intermittent Fasting
  Arms: Time-Restricted Feeding; Time-Restricted Feeding plus HMB

SUMMARY:
The objective of this study is to examine the effects of time-restricted feeding (TRF; consuming all calories within an 8-hour period of time each day) and resistance training, with or without the addition of the dietary supplement HMB, on body composition, muscular performance and physiological outcomes in active females.

ELIGIBILITY:
Inclusion Criteria:

* Female between 18 and 30 years of age
* Current university affiliation
* Weighing at least 110 pounds
* Generally healthy
* Resistance-trained
* Schedule availability to complete supervised resistance training
* Body fat percentage between 15 and 29%

Exclusion Criteria:

* Pregnant or trying to become pregnant
* Currently breastfeeding
* Any disease, condition or orthopedic limitation that would prevent safe participation in resistance training or time-restricted feeding
* Current smoker
* Presence of pacemaker or other electrical implant
* Allergic to dairy proteins

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Fat mass | 8 weeks
  Assessed using multi-compartment model
Fat-free mass | 8 weeks
  Assessed using multi-compartment model
Body fat percentage | 8 weeks
  Assessed using multi-compartment model
Upper body muscle hypertrophy | 8 weeks
  Muscle thickness of elbow flexor muscles
Lower body muscle hypertrophy | 8 weeks
  Muscle thickness of knee extensor muscles

SECONDARY OUTCOMES:
Lower body muscular strength | 8 weeks
  Assessed by 1RM on leg press
Lower body muscular power characteristics | 8 weeks
  Assessed during vertical jump and isometric squats
Lower body muscular endurance | 8 weeks
  Assessed by repetitions to failure on leg press
Upper body muscular strength | 8 weeks
  Assessed by 1RM on bench press
Upper body muscular endurance | 8 weeks
  Assessed by repetitions to failure on bench press
Cortisol awakening response | 8 weeks
  Assessed via analysis of saliva samples
Lipid panel | 8 weeks
  Measured from fasted blood sample
Blood glucose | 8 weeks
  Measured from fasted blood sample
Blood insulin | 8 weeks
  Measured from fasted blood sample
Blood C-reactive protein | 8 weeks
  Measured from fasted blood sample
Blood pressure | 8 weeks
  Measured using automated device
Arterial compliance | 8 weeks
  Assessed by applanation tonometry
Resting metabolic rate | 8 weeks
  Assessed by indirect calorimetry
Respiratory quotient | 8 weeks
  Assessed by indirect calorimetry
Mood | 8 weeks
  Assessed by questionnaire
Eating behavior | 8 weeks
  Assessed by three-factor eating questionnaire R18
Sleep quality | 8 weeks
  Assessed by Pittsburgh Sleep Quality Index
Physical activity level | 8 weeks
  Assessed by accelerometry.

CONTACTS AND LOCATIONS:
Overall Officials: Grant Tinsley, Ph.D., Principal Investigator — Texas Tech University
Locations (1):
- Texas Tech University, Lubbock, Texas, United States

REFERENCES:
- [Background] Moro T, Tinsley G, Bianco A, Marcolin G, Pacelli QF, Battaglia G, Palma A, Gentil P, Neri M, Paoli A. Effects of eight weeks of time-restricted feeding (16/8) on basal metabolism, maximal strength, body composition, inflammation, and cardiovascular risk factors in resistance-trained males. J Transl Med. 2016 Oct 13;14(1):290. doi: 10.1186/s12967-016-1044-0. PMID 27737674
- [Background] Tinsley GM, Forsse JS, Butler NK, Paoli A, Bane AA, La Bounty PM, Morgan GB, Grandjean PW. Time-restricted feeding in young men performing resistance training: A randomized controlled trial. Eur J Sport Sci. 2017 Mar;17(2):200-207. doi: 10.1080/17461391.2016.1223173. Epub 2016 Aug 22. PMID 27550719
- [Background] Tinsley GM, La Bounty PM. Effects of intermittent fasting on body composition and clinical health markers in humans. Nutr Rev. 2015 Oct;73(10):661-74. doi: 10.1093/nutrit/nuv041. Epub 2015 Sep 15. PMID 26374764
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717
- [Derived] Tinsley GM, Moore ML, Graybeal AJ, Paoli A, Kim Y, Gonzales JU, Harry JR, VanDusseldorp TA, Kennedy DN, Cruz MR. Time-restricted feeding plus resistance training in active females: a randomized trial. Am J Clin Nutr. 2019 Sep 1;110(3):628-640. doi: 10.1093/ajcn/nqz126. PMID 31268131